CLINICAL TRIAL: NCT05853198
Title: Circulating Tumor DNA as Surgical Biomarker in Patients With PancrEatic Adenocarcinoma for Statement of Resectability
Acronym: CASPER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3569
Record Dates: First submitted 2023-04-18; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: PDAC - Pancreatic Ductal Adenocarcinoma
Keywords: biomarker

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PDAC patients (Other): PDAC patients as described in the inclusion criteria
  Interventions: Other: ctDNA analysis

INTERVENTIONS:
Other: ctDNA analysis — ctDNA amount and mutations analysis

SUMMARY:
The main objective is the evaluation of the prognostic value of ctDNA (circulating tumor DNA) as a marker of surgical futility in patients with operable PDAC.

DETAILED DESCRIPTION:
In the era of personalized medicine and treatments guided by tumor biology, no specific tumor marker has real prognostic value. This is the reason why the search for a specific marker through a noninvasive blood test that can give indications on the usefulness of the resectability of pancreatic adenocarcinoma would be very valuable. Our project proposes the evaluation of ctDNA during various treatment courses of patients with PDAC in order to evaluate its efficacy as a prognostic and predictive marker of response to treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with PDAC with indication to surgical resection, including those undergoing upfront surgery or surgery following induction treatment. Non resectable patient defined as a patient with surgical indication at standard preoperative clinical, biological and morphological evaluation, but eventually not resected because of advanced disease or contraindications revealed during surgical exploration will be excluded
2. Non-metastatic status confirmed by an abdomen CT-scan (as our routine clinical practice).
3. Patients able to give a specific informed consent.
4. Age ≥ 18 years.

Exclusion Criteria:

1. Non resectable patient defined as a patient with surgical indication at standard preoperative clinical, biological and morphological evaluation, but eventually not resected because of advanced disease or contraindications revealed during surgical exploration will be excluded (drop-out)
2. Non-controlled congestive heart failure.
3. Non-treated angina.
4. Recent myocardial infarction (in the previous year).
5. Non-controlled AHT (SBP >160 mm or DBP > 100 mm, despite optimal drug treatment).
6. Long QT.
7. Major non-controlled infection.
8. Severe liver failure.
9. Age < 18 years.
10. Informed consent not signed.
11. Pregnant or breastfeeding women and women of child-bearing age not using effective means of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2022-12-29 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Disease relapse | 2 years
  disease relapse at 2 years after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- AOUI Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: Undecided